CLINICAL TRIAL: NCT01120600
Title: A Phase III Randomized, Placebo-Controlled Clinical Trial to Assess the Safety and Efficacy of Odanacatib (MK-0822) in the Treatment of Men With Osteoporosis Treated With Vitamin D and Calcium
Brief Title: A Study to Assess Safety and Efficacy of Odanacatib (MK-0822) in Men With Osteoporosis (MK-0822-053)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0822-053; 2010_532 (Other: Merck)
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — odanacatib; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Odanacatib 50 mg once weekly (Experimental): Participants will receive one Odanacatib 50 mg tablet once weekly. In addition, they will receive a weekly dose 5600 IU of open-label Vitamin D3 as well as a sufficient supply of open-label calcium carbonate so that their total daily calcium intake from both dietary and supplemental sources is approximately 1200 mg.
  Interventions: Drug: Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Placebo once weekly (Placebo Comparator): Participants will receive one Placebo tablet once weekly. In addition, they will receive a weekly dose 5600 IU of open-label Vitamin D3 as well as a sufficient supply of open-label calcium carbonate so that their total daily calcium intake from both dietary and supplemental sources is approximately 1200 mg.
  Interventions: Drug: Placebo for Odanacatib; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Drug: Odanacatib — One 50 mg tablet once weekly
  Other Names: MK-0822
  Arms: Odanacatib 50 mg once weekly
Drug: Placebo for Odanacatib — One 50 mg tablet once weekly
  Arms: Placebo once weekly
Dietary Supplement: Vitamin D3 — 5600 IU of open-label Vitamin D3 once weekly
Dietary Supplement: Calcium carbonate — Sufficient amount of open-label calcium carbonate so that daily calcium intake from both dietary and supplementary sources in approximately 1200 mg

SUMMARY:
The purpose of this study is to test the hypothesis that treatment with odanacatib will result in increased bone mineral density (BMD) compared to treatment with placebo. This study will also evaluate the safety and efficacy of odanacatib for male osteoporosis participants.

DETAILED DESCRIPTION:
The original study was divided into two parts, with the primary analysis of endpoints to occur at 24 months and participants will then remain in the study for an additional 12 months (Part 2). Amendment 1 of the protocol removed the additional 12 month period and the Month 36 BMD analysis was deleted.

ELIGIBILITY:
Inclusion Criteria:

* Is a male between 40 and 95 years of age
* Has osteoporosis
* Has anatomy suitable for dual energy x-ray absorptiometry (DXA) scan of the lumbar spine and and hip
* Is ambulatory

Exclusion Criteria:

* Is currently on oral bisphosphonates or other treatment for osteoporosis
* Had previous hip fragility fracture and is a candidate for standard of care therapy
* Has had a fragility fracture (vertebral or non-vertebral fractures indicating reduced bone strength) within 12 months
* Has had more then one previous vertebral fracture
* Has been diagnosed with metabolic bone disorder other than osteoporosis
* Is Vitamin D deficient
* Has a history of renal stones
* Has active parathyroid disease
* Has history of thyroid disease not well controlled by medication
* Is diagnosed with secondary osteoporosis
* Has a daily calcium intake of <1,200 mg and is unwilling to take study prescribed supplements or increase dietary intake, such that his daily calcium intake is at least 1200 mg
* Has a history of malignancy ≤5 years prior to signing informed consent
* Has been diagnosed with hypogonadism due to causes that affect multiple organ and body systems

Ages: 40 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 294 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2013-07-22 (Actual); Study Completion 2013-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Binkley N, Orwoll E, Chapurlat R, Langdahl BL, Scott BB, Giezek H, Santora AC. Randomized, controlled trial to assess the safety and efficacy of odanacatib in the treatment of men with osteoporosis. Osteoporos Int. 2021 Jan;32(1):173-184. doi: 10.1007/s00198-020-05701-9. Epub 2020 Nov 17. PMID 33200257

RESULTS

PARTICIPANT FLOW:
Groups:
- Odanacatib 50 mg Once Weekly: Participants received one Odanacatib 50 mg tablet once weekly. In addition, they received a weekly dose 5600 IU of open-label Vitamin D3 as well as a sufficient supply of open-label calcium carbonate so that their total daily calcium intake from both dietary and supplemental sources was approximately 1200 mg.
- Placebo Once Weekly: Participants received one Placebo tablet once weekly. In addition, they received a weekly dose 5600 IU of open-label Vitamin D3 as well as a sufficient supply of open-label calcium carbonate so that their total daily calcium intake from both dietary and supplemental sources was approximately 1200 mg.
Period: Overall Study
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Started | 147 | 147
Treated | 146 | 146
Completed | 128 | 115
Not Completed | 19 | 32
Not completed — Adverse Event | 7 | 7
Not completed — Excessive Bone Loss | 0 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.2) | 68.7 (7.7) | 68.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 147 | 147 | 294

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Month 24
Description: Lumbar spine BMD was assessed by dual energy X-ray absorptiometry (DXA) at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who took at least one dose of blinded study treatment and had available lumbar spine BMD data for Baseline and Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 112 | 107
Percentage change | 6.86 [6.08 to 7.64] | 1.27 [0.48 to 2.06]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; A constrained full likelihood longitudinal data analysis (cLDA) method was used for this statistical analysis. The cLDA model included the baseline measurement and all post-baseline percent changes from baseline in the response vector, with fixed effects for treatment, time, geographic region, machine type and treatment-by-time interaction, geographic region-by-time interaction, and machine type-by-time interaction; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = 5.59, 95% CI 2-sided [4.48 to 6.7]

2. Secondary Outcome: Percentage Change From Baseline in Total Hip BMD at Month 24
Description: Total hip BMD was assessed by DXA at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who took at least one dose of blinded study treatment and had available total hip BMD data for Baseline and Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 111 | 105
Percentage change | 1.91 [1.38 to 2.43] | -0.11 [-0.65 to 0.42]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; A cLDA method was used for this statistical analysis. The cLDA model included the baseline measurement and all post-baseline percent changes from baseline in the response vector, with fixed effects for treatment, time, geographic region, machine type and treatment-by-time interaction, geographic region-by-time interaction, and machine type-by-time interaction; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = 2.02, 95% CI 2-sided [1.27 to 2.77]

3. Secondary Outcome: Percentage Change From Baseline in Femoral Neck BMD at Month 24
Description: Femoral Neck BMD was assessed by DXA at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who took at least one dose of blinded study treatment and had available femoral neck BMD data for Baseline and Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 111 | 105
Percentage change | 1.69 [0.82 to 2.55] | 0 [-0.89 to 0.88]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.008, cLDA; Difference in Least Squares Means = 1.69, 95% CI 2-sided [0.45 to 2.93]

4. Secondary Outcome: Percentage Change From Baseline in Trochanter BMD at Month 24
Description: Trochanter BMD was assessed by DXA at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who took at least one dose of blinded study treatment and had available trochanter BMD data for Baseline and Month 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 111 | 105
Percentage change | 2.77 [1.94 to 3.6] | 0.66 [-0.18 to 1.5]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = 2.12, 95% CI 2-sided [0.93 to 3.3]

5. Secondary Outcome: Percentage Change From Baseline in Serum C-Telopeptides of Type 1 Collagen (s-CTx) at Month 24
Description: Serum samples were collected to evaluate biochemical markers for s-CTx, which were measured at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who had no important deviations from the protocol that may have substantially affected the results, and had available s-CTx data for Baseline and Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 112 | 102
Percentage change | -20.07 [-28.36 to -10.82] | 56.51 [40.01 to 74.96]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = -76.58, 95% CI 2-sided [-92.56 to -60.61]

6. Secondary Outcome: Percentage Change From Baseline in Urine Collagen N-Telopeptide/Creatinine Ratio (U-NTx/Cr) at Month 24
Description: Urine samples were collected to evaluate biochemical markers for u-NTx/Cr, which were measured at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who had no important deviations from the protocol that may have substantially affected the results, and had available U-NTx/Cr data for Baseline and Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 111 | 102
Percentage change | -61.43 [-64.71 to -57.85] | 6.65 [-2.68 to 16.87]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, cLDA; Difference in Least Squares Means = -68.08, 95% CI 2-sided [-78.1 to -58.06]

7. Secondary Outcome: Percentage Change From Baseline in Serum Bone-Specific Alkaline Phosphatase (s-BSAP) at Month 24
Description: Serum samples were collected to evaluate biochemical markers for s-BSAP, which were measured at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who had no important deviations from the protocol that may have substantially affected the results, and had available s-BSAP data for Baseline and Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 114 | 110
Percentage change | -5.28 [-9.76 to -0.57] | 2.66 [-2.25 to 7.82]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.019, cLDA; Difference in Least Squares Means = -7.94, 95% CI 2-sided [-14.58 to -1.31]

8. Secondary Outcome: Percentage Change From Baseline in Serum N-Terminal Propeptides of Type I Collagen (s-P1NP) at Month 24
Description: Serum samples were collected to evaluate biochemical markers for s-P1NP, which were measured at Baseline and at Month 24.
Time Frame: Baseline and Month 24
Population: All randomized participants who had no important deviations from the protocol that may have substantially affected the results, and had available s-P1NP data for Baseline and Week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 114 | 100
Percentage change | -10.94 [-17.27 to -4.14] | 5.06 [-2.47 to 13.17]
Statistical Analysis 1: Comparison: Odanacatib 50 mg Once Weekly vs Placebo Once Weekly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.001, cLDA; Difference in Least Squares Means = -16, 95% CI 2-sided [-25.74 to -6.27]

9. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not it is considered related to the study drug.
Time Frame: Up to 24 months (plus 14 days) after first dose of study drug
Population: All randomized participants who took at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 146 | 146
Participants | 113 | 114

10. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 9
Time Frame: Up to 24 months after first dose of study drug
Population: All randomized participants who took at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Number analyzed (Participants) | 146 | 146
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: Up to 24 months (plus 14 days) after first dose of study drug
Description: All randomized participants who took at least one dose of study drug
Arm/Group | Odanacatib 50 mg Once Weekly | Placebo Once Weekly
Serious Adverse Events (participants affected / at risk) | 24/146 | 24/146
Other Adverse Events (participants affected / at risk) | 30/146 | 44/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odanacatib 50 mg Once Weekly (N=146) | Placebo Once Weekly (N=146)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Retroperitoneal infection (Infections and infestations) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (4)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Odanacatib 50 mg Once Weekly (N=146) | Placebo Once Weekly (N=146)
Influenza like illness (General disorders) | 4 (4) | 9 (11)
Nasopharyngitis (Infections and infestations) | 14 (18) | 15 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 10 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 12 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.